CLINICAL TRIAL: NCT04710719
Title: Efficacy of Post-Surgical Intralesional Injection With Triamcinolone Versus Triamcinolone Plus Fluorouracil in the Treatment of Keloids
Brief Title: Post-Surgical Injection With Triamcinolone Versus Triamcinolone/Fluorouracil in Treatment of Keloids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Our Lady of the Lake Hospital (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Keloid_5FU/TAC
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Keloid; Keloid Scar Following Surgery
MeSH Terms: conditions — Keloid | interventions — Triamcinolone; Fluorouracil

STUDY DESIGN:
Intervention Model Description: 2 cohort arms, single blinded; 1=TAC alone, 2=TAC+5FU
Who Masked: Participant
Masking Description: Participants will not be aware of which injection they will be receiving in follow up treatment for their keloid (TAC alone or TAC/5FU)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAC only (Active Comparator): Participants will be treated with adjuvant intralesional TAC 40mg/mL 7-10 days post-op and then every 4 weeks for a total of 3 injections. Assessments will be performed at 3, 6, 9, and 12 months after completion of treatment. At each time point, a member of the study team and patient will complete their respective portion of the Patient and Observer Scar Assessment Scale (POSAS).
  Interventions: Drug: Triamcinolone Injection
- TAC + 5FU (Active Comparator): Participants will be treated with adjuvant intralesional TAC and 5FU at a dose of 0.1mg TAC for every 0.9mg 5FU 7-10 days post-op then every 4 weeks for a total of 3 injections. Assessments will be performed at 3, 6, 9, and 12 months after completion of treatment. At each time point, a member of the study team and patient will complete their respective portion of the Patient and Observer Scar Assessment Scale (POSAS).
  Interventions: Drug: Triamcinolone Injection and 5-fluorouracil injection

INTERVENTIONS:
Drug: Triamcinolone Injection — Post surgical injection at site of keloid with TAC for 3 injections
  Other Names: TAC
  Arms: TAC only
Drug: Triamcinolone Injection and 5-fluorouracil injection — Post surgical injection at site of keloid with TAC and 5FU for 3 injections
  Other Names: TAC + 5FU
  Arms: TAC + 5FU

SUMMARY:
There have been many modalities utilized in the treatment of keloids of the head and neck, however none have been universally successful. The most widely utilized non-surgical intervention is primary intralesional injection with triamcinolone (TAC) which inhibits the proliferation of fibroblasts, inhibits collagen synthesis, and increases collagenase production, or fluorouracil (5-FU), a potent inhibitor of fibroblast proliferation. Despite the abundance of studies evaluating primary intralesional injection for keloids, there are limited studies available regarding the efficacy of primary surgical excision followed by adjuvant intralesional injection. The proposed study herein would serve to improve the level of evidence and to establish the safety and efficacy of combined intralesional TAC+5FU for keloids following surgical excision.

DETAILED DESCRIPTION:
This is a single blinded, prospective randomized controlled trial of patients who elect for surgical treatment of keloids at the Center for Facial Plastic and Reconstructive Surgery at Our Lady of the Lake Regional Medical Center (OLOLRMC), a tertiary referral center affiliated with the Louisiana State University Health Sciences Center (LSUHSC) teaching system. Power analysis estimated approximately 134 patients total (67 per group) for 80% power to detect a difference at the 5% confidence level. This is based off of a prior group's study comparing primary intralesional injection with TAC vs TAC+5FU (no surgery). That study showed 39.2% recurrence with TAC vs 17.5% with TAC+5FU.

The patients enrolled in the study will be randomized to one of two arms: surgical excision+TAC or surgical excision+TAC+5FU. Randomization will be performed using a permuted block randomization algorithm (Ex. AABBABABABBABBAA, where A=TAC only group and B=TAC +5FU). All patients will undergo surgical excision of the keloid, either under general anesthesia in the operating room or local anesthesia in the clinic setting depending on patient age and preference. The goal of excision will be complete extra-lesional excision with primary closure. It will be noted if a patient requires intra-lesional excision or additional reconstructive techniques such as advancement flap, skin grafting, or allografting (i.e. Integra). Monofilament sutures will be used preferentially to prevent local inflammatory reaction which can precipitate keloid formation. In group 1 (surgical excision+TAC), all patients will be treated with adjuvant intralesional TAC 40mg/mL 7-10 days post-op and then every 4 weeks for a total of 3 injections. The triamcinolone vial will be obtained from pharmacy and drawn up by the physician prior to injection. In group 2 (surgical excision+TAC+5FU), all patients will be treated with adjuvant intralesional TAC and 5FU at a dose of 0.1mg TAC for every 0.9mg 5FU 7-10 days post-op then every 4 weeks for a total of 3 injections. The mixture of TAC+5FU will be prepared by the pharmacy and delivered to the physician prior to injection. The goal volume of injection for both arms of the study will be 0.1cc per cm2 of scar excised, though any deviations from this and the rationale will be noted.

Assessments will be performed at 3, 6, 9, and 12 months after completion of treatment. At each time point, a member of the study team and patient will complete their respective portion of the Patient and Observer Scar Assessment Scale (POSAS) which has been proven as a reliable and valid method of assessing keloid scars (5). The observer portion of the survey to be completed by the study team assesses vascularity, pigmentation, thickness, pliability, and surface area of the lesion. The patient portion of the survey focuses on the overall cosmetic and functional sequela including pain, itching, color, stiffness, thickness, and irregularity. Patients will also be asked about any side effects experienced. Each portion of the POSAS will be blinded from the study team member and the participant until both have completed the survey at each visit, so that one set of answers will not bias the other. If a patient demonstrates signs of recurrence or return of symptoms, there will be the option for additional injections within the patient's originally designated study arm. However, if early analysis demonstrates the alternative study arm to have superior efficacy, there will be the option to continue injections with the alternative study arm injection.

Data collection will include demographic data such as age, gender, race, and Fitzpatrick skin type, as well as location of the keloid, etiology (trauma, post-surgical, etc.), and prior treatments if any. The size and thickness of each lesion, secondary defect size following adjacent tissue transfer, and amount of adjuvant medication injected during each adjuvant injection will be collected. Data analysis will include overall efficacy as well as stratification by variables such as the location of the lesion, size of the lesion, and prior treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any age
* Subjects with at least one keloid of any size located in the head and neck region

Exclusion Criteria:

* subjects with comorbidities prohibiting local injection of either TAC or 5FU including pregnancy, lactation, or planning pregnancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Keloid Recurrence by visual assessment meaning either there is or is not a keloid physically present (determined by number of keloids observed and rate of recurrence after treatment) | 12 months
  Treatment effective if no keloid recurrence is visible by 12 months post treatment

SECONDARY OUTCOMES:
Symptomatology-assessed by Patient and Observer Scar Assessment Scale | 3 months
  Effectiveness of treatment on symptoms (pruritus, pain, hyperpigmentation or other side effects) as determined by changes in the POSAS survey (1 being "not observed" to 10 being "present always" and also by visual assessment by the physician

CONTACTS AND LOCATIONS:
Overall Officials: Justin Sowder, MD, Principal Investigator — Louisiana State University Health Sciences Center - New Orleans
Locations (1):
- Our Lady of the Lake Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ren Y, Zhou X, Wei Z, Lin W, Fan B, Feng S. Efficacy and safety of triamcinolone acetonide alone and in combination with 5-fluorouracil for treating hypertrophic scars and keloids: a systematic review and meta-analysis. Int Wound J. 2017 Jun;14(3):480-487. doi: 10.1111/iwj.12629. Epub 2016 Jul 18. PMID 27427423
- [Background] Khalid FA, Mehrose MY, Saleem M, Yousaf MA, Mujahid AM, Rehman SU, Ahmad S, Tarar MN. Comparison of efficacy and safety of intralesional triamcinolone and combination of triamcinolone with 5-fluorouracil in the treatment of keloids and hypertrophic scars: Randomised control trial. Burns. 2019 Feb;45(1):69-75. doi: 10.1016/j.burns.2018.08.011. Epub 2018 Oct 16. PMID 30340861
- [Background] Al-Attar A, Mess S, Thomassen JM, Kauffman CL, Davison SP. Keloid pathogenesis and treatment. Plast Reconstr Surg. 2006 Jan;117(1):286-300. doi: 10.1097/01.prs.0000195073.73580.46. PMID 16404281
- [Background] Davison SP, Dayan JH, Clemens MW, Sonni S, Wang A, Crane A. Efficacy of intralesional 5-fluorouracil and triamcinolone in the treatment of keloids. Aesthet Surg J. 2009 Jan-Feb;29(1):40-6. doi: 10.1016/j.asj.2008.11.006. PMID 19233005
- [Background] Wu XL, Gao Z, Song N, Liu W. [Clinical study of auricular keloid treatment with both surgical excision and intralesional injection of low-dose 5-fluorouracil and corticosteroids]. Zhonghua Yi Xue Za Zhi. 2009 Apr 28;89(16):1102-5. Chinese. PMID 19595138
- [Background] Nicholas RS, Falvey H, Lemonas P, Damodaran G, Ghannem A, Selim F, Navsaria H, Myers S. Patient-related keloid scar assessment and outcome measures. Plast Reconstr Surg. 2012 Mar;129(3):648-656. doi: 10.1097/PRS.0b013e3182402c51. PMID 22373972